CLINICAL TRIAL: NCT06151847
Title: Reduced Dose Fludarabine/Cyclophosphamide Lymphodepletion Before Tumor-Infiltrating Lymphocyte Therapy With Lifileucel in Metastatic Melanoma
Brief Title: Lifileucel With Reduced Dose Fludarabine/Cyclophosphamide Lymphodepletion and Interleukin-2 for the Treatment of Patients With Unresectable or Metastatic Melanoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Iovance Biotherapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, Muhammad Mushtaq, Assistant Professor, University of Kansas Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00150697; NCI-2023-09309 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IIT-2022-LDTIL; STUDY00150697 (Other: University of Kansas Cancer Center); P30CA168524 (NIH)
Record Dates: First submitted 2023-11-17; First posted 2023-11-30 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Clinical Stage IV Cutaneous Melanoma AJCC v8; Metastatic Melanoma; Pathologic Stage IIIC Cutaneous Melanoma AJCC v8; Unresectable Melanoma
MeSH Terms: conditions — Melanoma | interventions — Specimen Handling; Cyclophosphamide; fludarabine; Interleukin-2; 4-toluenesulfonyl fluoride; lifileucel; Magnetic Resonance Spectroscopy; Transurethral Resection of Bladder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Lifileucel) (Experimental): Lifileucel (LN-144) is an autologous Tumor Infiltrating Lymphocytes (TIL) cell therapy. A tumor sample is resected from each patient for lifileucel manufacturing. Patients then receive the lifileucel regimen which consists of a reduced dose non-myeloablative lymphodepletion, lifileucel infusion followed by interleukin-2.
  Interventions: Procedure: Biospecimen Collection; Drug: Cyclophosphamide; Procedure: Echocardiography; Drug: Fludarabine; Biological: Interleukin-2; Biological: Lifileucel; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Procedure: Tumor Resection

INTERVENTIONS:
Procedure: Biospecimen Collection — A tumor sample is resected from each patient and cultured ex vivo to expand the population of tumor infiltrating lymphocytes. After lymphodepletion, patients are infused with Lifileucel followed by IL-2
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection; Undergo blood sample collection
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B-518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719; WR-138719
Procedure: Echocardiography — Undergo echocardiography
  Other Names: EC
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Biological: Interleukin-2 — Given IV
  Other Names: Epidermal Thymocyte Activating Factor; ETAF; hIL-2; IL-2; IL2; IL2 Protein; Interleukin 2; Interleukin 2 Precursor; Interleukin II; Lymphocyte Mitogenic Factor; Mitogenic Factor; Ro-236019; T Cell Growth Factor; T-Cell Growth Factor; TCGF; Thymocyte Stimulating Factor; TSF
Biological: Lifileucel — Given IV
  Other Names: Autologous TIL LN-144; Autologous Tumor Infiltrating Lymphocytes LN-144; Contego; Lifileuecel; LN-144
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Multigated Acquisition Scan — Undergo MUGA scan
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Procedure: Tumor Resection — Undergo tumor resection

SUMMARY:
This phase II trial tests how well lifileucel, with reduce dose fludarabine and cyclophosphamide for lymphodepletion and interleukin-2, work for treating patients with melanoma that cannot be removed by surgery (unresectable) or that has spread from where it first started (primary site) to other places in the body (metastatic).Lifileucel is made up of specialized immune cells called lymphocytes or T cells that are taken from a patient's tumor, grown in a manufacturing facility and infused back into the preconditioned patient to attack the tumor. Giving Lifileucel with a reduced dose of fludarabine and cyclophosphamide for lymphodepletion and interleukin -2 is being studied in patients with unresectable or metastatic melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. The percentage of total TIL clones as measured by the T-cell receptor (TCR) population shared between the tumor infiltrating lymphocyte (TIL) product and peripheral blood mononuclear cells (PBMC).

SECONDARY OBJECTIVES:

I. To evaluate the efficacy parameters of lifileucel (LN-144) in combination with a reduced dose lymphodepletion in patients with unresectable or metastatic melanoma by assessing objective response rate (ORR), progression-free survival (PFS), and overall survival (OS).

II. To characterize the safety profile of lifileucel (LN-144) in combination with a reduced dose lymphodepletion regimen in patients with unresectable or metastatic melanoma.

EXPLORATORY OBJECTIVE:

I. Blood and tumor samples will be banked for future correlative analyses, including flow cytometry, next generation sequencing, immunogenomics and RNA sequencing to characterize the immunome and microenvironment.

OUTLINE:

Patients undergo tumor resection surgery. After the lifileucel is manufactured (approximately 4 weeks later), patients receive cyclophosphamide intravenously (IV) on days -4 to -2 and fludarabine IV on days -4 to -1. Patients then receive lifileucel IV on day 0. Patients also receive up to 6 doses of intraleukin-2 IV.

After completion of study treatment, patients are followed up at day 28, 42, 84, 126, 180, 365, month 18, and month 24.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age ≥ 18 years Enrollment of patients ≥ 70 years of age may be allowed at principal investigator discretion.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 1
* At least one measurable target lesion, as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1

  * Lesions in previously irradiated areas (or other local therapy) should not be selected as target lesions, unless treatment was ≥ 3 months prior to Screening, and there has been demonstrated disease progression in that lesion
* Women of childbearing potential must have a negative serum pregnancy test 48 hours prior to initiating treatment
* Patients with unresectable or metastatic melanoma (stage IIIc or stage IV)
* Patients must have progressed following 1-3 prior systemic therapy including a programmed cell death protein-1 (PD-1) blocking antibody; and if proto-oncogene B-Raf (BRAF) V600 mutation positive, a BRAF inhibitor or BRAF inhibitor in combination mitogen-activated extracellular signal-regulated kinase (MEK) inhibitor
* At least one resectable lesion (or aggregate of lesions resected) of a minimum 1.5 cm in diameter post-resection to generate TIL; surgical removal with minimal morbidity (defined as any procedure for which expected hospitalization is ≤ 3 days)
* Adequate hematologic and organ function
* Patients must have recovered from all prior therapy-related adverse events (AEs) to ≤ grade 1 (per Common Terminology Criteria for Adverse Events [CTCAE] version [v] 5.0), except for alopecia or vitiligo, prior to enrollment (tumor resection)

  * Patients with documented ≥ grade 2 diarrhea or colitis because of previous treatment with immune checkpoint inhibitor(s) must have been asymptomatic for at least 6 months and/or had a normal colonoscopy post-immune checkpoint inhibitor treatment, by visual assessment, prior to tumor resection
* Patients with immunotherapy-related endocrinopathies stable for at least 6 weeks (eg, hypothyroidism), and controlled with hormonal replacement (non-corticosteroids), are allowed
* Patients must have a washout period of ≥ 28 days from prior anticancer therapy(ies) to the start of the planned reduced dose lymphodepletion (RDL) preconditioning regimen:

  * Targeted therapy: MEK/BRAF or other targeted agents
  * Chemotherapy
  * Immunotherapy: anti-CTLA-4/anti-PD-1, other monoclonal antibodies (mAb), or vaccine
  * Palliative radiation therapy is permitted so long as it does not involve lesions being selected for TIL, or as target or non-target lesions. Washout is not required if all related toxicities have resolved to ≤ grade 1 as per CTCAE v 5.0
* Women of child-bearing potential and men with partners of child-bearing potential must agree to practice sexual abstinence or to use the forms of contraception listed in Child-Bearing Potential/Pregnancy section for the duration of study participation and for 12 months following the last dose of IL-2 or until the first dose of the next anti-cancer therapy, whichever occurs first

Exclusion Criteria:

* Current or anticipating use of other anti-neoplastic or investigational agents while participating in this study
* Is pregnant or breastfeeding
* Patients who have active medical illness(es) that would pose increased risk for study participation, including active systemic infections requiring systemic antibiotics, coagulation disorders, or other active major medical illnesses of the cardiovascular, respiratory, or immune system
* Patients who have been shown to be BRAF mutation positive (V600), but have not received prior systemic therapy with a BRAF inhibitor alone or a BRAF inhibitor in combination with a MEK inhibitor
* Patients who have received an organ allograft or prior cell transfer therapy
* Patients with melanoma of uveal/ocular origin
* Patients who have a history of hypersensitivity to any component or excipient of Lifileucel or other study drugs
* Patients who have any form of primary immunodeficiency (such as severe combined immunodeficiency disease [SCID] and acquired immunodeficiency syndrome [AIDS])
* Patients who have a left ventricular ejection fraction (LVEF) < 45% or New York Heart Association (NYHA) functional classification class > 1
* Patients who have a documented forced expiratory volume in 1 second (FEV1) of ≤ 60%
* Patients who have had another primary malignancy within the previous 3 years (except for carcinoma in situ of the breast, cervix, or bladder; localized prostate cancer; and non-melanoma skin cancer that has been adequately treated)
* Patients with symptomatic and/or untreated brain metastases (of any size and any number)

  * Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-12-21 (Actual); Primary Completion 2025-11-27 (Estimated); Study Completion 2025-11-27 (Estimated)

PRIMARY OUTCOMES:
Percentage of total T-cell receptor (TCR) populations shared between the TIL product and peripheral blood mononuclear cells (PBMCs) | At day + 42
  The TCR population is calculated as the frequencies of unique CDR3 sequences as measured by HTBIvc assay. Will be summarized with respect to mean and standard deviation. The percentage changes will also be presented with respect to visual diagrams for each person, e.g., waterfall plot

SECONDARY OUTCOMES:
Safety: Incidence of treatment emergent adverse events | From start of treatment to 6 months after TIL
  Defined as all grades and any attribution until day 28 (EOT visit) after infusion, grade 3-4 of any attribution from day 28 to 6 months, only grade 3-4 attributed to study drugs after 6 months evaluated by Common Terminology Criteria in Adverse Events (CTCAE). Will be presented as percentage with 95% confidence intervals and tabulated by type and grade.
Safety: Incidence of serious adverse events | From start of treatment to 6 months after TIL
  Defined as all grades and any attribution until day 28 (EOT visit) after infusion, grade 3-4 of any attribution from day 28 to 6 months, only grade 3-4 attributed to study drugs after 6 months evaluated by CTCAE. Will be presented as percentage with 95% confidence intervals and tabulated by type and grade.
Transfusion requirements | From start of treatment to 6 months after TIL
  Defined as all grades and any attribution until day 28 (EOT visit) after infusion, grade 3-4 of any attribution from day 28 to 6 months, only grade 3-4 attributed to study drugs after 6 months evaluated by CTCAE. Will be presented as percentage with 95% confidence intervals and will be summarized with respect to mean and standard deviation.
Length of hospital stay | From start of treatment to 6 months after TIL
  Defined as all grades and any attribution until day 28 (EOT visit) after infusion, grade 3-4 of any attribution from day 28 to 6 months, only grade 3-4 attributed to study drugs after 6 months evaluated by CTCAE. Will be presented as percentage with 95% confidence intervals and will be summarized with respect to mean and standard deviation.
Overall response rate | From start of treatment until the end of treatment, up to 2 years
  Measured by Response Evaluation Criteria in Solid Tumor (RECIST) 1.1. Will be presented as percentage with 95% confidence internal using Clopper-Pearson Exact method.
Progression free survival | From start of treatment until objective tumor progression or death, up to 2 years
  Will be summarized with Kaplan-Meir curves and estimation of medians with 95% confidence intervals.
Overall survival | From start of treatment to death due to any cause, up to 2 years
  Will be summarized with Kaplan-Meir curves and estimation of medians with 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Umair Mushtaq, Principal Investigator — University of Kansas
Locations (1):
- University of Kansas Cancer Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Mushtaq MU, Abdelhakim H, Selby L, Shahzad M, Abhyankar SH, McGuirk JP, Doolittle GC. Reduced dose fludarabine and cyclophosphamide lymphodepletion before tumor-infiltrating lymphocyte therapy in melanoma. Future Oncol. 2025 Jun;21(13):1631-1637. doi: 10.1080/14796694.2025.2498842. Epub 2025 May 9. PMID 40343719